CLINICAL TRIAL: NCT00386178
Title: Comparison of Gamma-tocopherol Supplementation in Allergic Asthmatics and Normal Volunteers
Brief Title: Safety Study of a Vitamin E Supplement in Normal Volunteers and Those With Both Allergy and Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: David Peden, MD/Principal Investigator, UNC Center for Environmental Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 05-2833
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Asthma
Keywords: vitamin E; gamma tocopherol; moderate to severe asthma; healthy subjects
MeSH Terms: conditions — Asthma | interventions — gamma-Tocopherol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Vitamin E supplement rich in gamma tocopherol
  Interventions: Drug: Vitamin E supplement rich in gamma tocopherol

INTERVENTIONS:
Drug: Vitamin E supplement rich in gamma tocopherol — daily dose of Vitamin E supplement rich in gamma tocopherol
  Other Names: Maxi-Gamma

SUMMARY:
Gamma tocopherol (gt) is a naturally occurring form of vitamin E that is found in many foods, and is also commercially available as a vitamin supplement. The purpose of this Phase 1 research study is to see if two doses of gt, 600mg and 1200mg, are safe (do not cause gastrointestinal distress or other problems), and can cause changes in your blood levels of gt and other antioxidants. This study will also examine if there is a difference in response between asthmatic and non-asthmatic adults when taking the same dose of gt. Phase 1 research studies like this one are not intended to be a treatment, but are a scientific investigation.

DETAILED DESCRIPTION:
This is designed as an open label study of the effect of 600 mg and 1200mg gamma tocopherol (gt), orally administered daily for 8 days, on serum antioxidant levels in asthmatics and healthy volunteers. Each course of gamma tocopherol will be followed by a 7-8 day wash out period and serum testing to ensure that blood levels are back to baseline prior to starting the next course. The gamma tocopherol will be obtained from Yasoo Health Inc and contains 623mg gt per 830 mg gelatin capsule.

Allergy skin testing to a battery of allergens common to the region will be performed to determine the state of atopy both prior to drug administration and after the 8 day course. Allergic volunteers will be asked to abstain from taking any antihistamines during the 3 days prior to the skin testing. Repeat allergy testing will not be performed on subjects unable to hold antihistamines for health reasons, or on non-allergic volunteers who demonstrate no response to baseline testing. Spirometry will be performed to determine the current level of lung function. Subjects will be asked to refrain from taking vitamin supplements, non-steroidal anti-inflammatory medications and other dietary supplements.

ELIGIBILITY:
Inclusion Criteria: allergic asthmatic cohort

* Specific allergy to at least one of the following allergen preparations: (House Dust Mite f, House dust mite p, Cockroach, Tree mix, Grass Mix, Weed Mix, Mold Mix 1, Mold Mix 2, Rat, Mouse, Guinea Pig, Rabbit, Cat or Dog) confirmed by positive immediate skin test response.
* Oxygen saturation of > 94 % at baseline
* Blood pressure within the following parameters (Systolic between 150 - 90,Diastolic between 100-60 mm Hg)
* Moderate or severe persistent asthma according to NHLBI definitions including history of one of the following: 1)Episodic wheezing, chest tightness or shortness of breath consistent with asthma occurring at least once a week that may affect activity;2)Asthma symptoms occurring at night or during sleep at least 1 time per week; 3)measured FEV1 or FVC is <80% of predicted; OR 4)physician diagnosed moderate or severe persistent asthma which is currently treated or controlled with maintenance medication including moderate or high dose inhaled corticosteroid, or any dose of inhaled corticosteroid and a long-acting inhaled B2-agonist

Inclusion Criteria- healthy volunteer cohort

* Oxygen saturation > 94 % at baseline
* Blood pressure within the following parameters (Systolic between 150 - 90, Diastolic between 100-60 mm Hg)
* No active allergies
* No physician diagnosis of asthma since age 6

Exclusion Criteria:

* Any chronic medical condition considered by the PI as a contraindication to receiving gamma tocopherol, including significant cardiovascular disease, diabetes requiring medication, chronic renal disease, chronic thyroid disease, kidney disease or coagulation defects.
* Use of inhaled steroids, cromolyn or leukotriene inhibitors (montelukast or zafirlukast) which have been used for at least one month are allowed. Patients must be on a stable regimen of maintenance asthma therapy which has not changed in the past month prior to entrance into the study.
* NSAID or ASA use within 48 hours of beginning the study, and inability to suspended use of these medications during the length of the study.
* Use of anticoagulants including warfarin, heparin, or clopidogrel.
* Diagnosis of anemia or abnormal blood counts at screening
* Pregnancy or nursing a baby. As this is a phase I study, the potential risk to a fetus cannot be justified.
* Children will not be included in this study as the potential risk to a growing child cannot be justified.
* Adults age 51 and older are excluded as the potential for concomitant illness in this population increases the risk for confounding the data.
* Known vagal response to venipuncture
* Abnormal PT or PTT values at screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
serum levels of gamma tocopherol and its metabolites after eight days of supplementation | eight days

SECONDARY OUTCOMES:
latency between the first dose and peak levels of gamma tocopherol | levels at points within 24 hours
effect of gamma tocopherol supplementation on other antioxidants | 8 days
effect of supplementation with gamma tocopherol on changes on cell surface marker expression on circulating monocytes and macrophages and on these cells' response to ex vivo LPS challenge | 1-8 days

CONTACTS AND LOCATIONS:
Overall Officials: David B Peden, MD, MS, Principal Investigator — University of North Carolina at Chapel Hill, Dept of Pediatrics / Center for Environmental Medicine, Asthma and Lung Biology
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology at the University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Center for Environmental Medicine, Asthma and Lung Biology — http://www.med.unc.edu/cemalb